CLINICAL TRIAL: NCT00793845
Title: Tandem High-dose Chemotherapy and Autologous Stem Cell Rescue in Patients With High-risk Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-07-002
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Neuroblastoma
Keywords: tandem high-dose chemotherapy for high-risk neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Cyclophosphamide; Etoposide; Carboplatin; Thiotepa; Melphalan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High risk neuroblastoma (Experimental): 1. Conventional chemotherapy (9 cycles)
  2. Surgery conventional chemotherapy (after 6 cycles of chemotherapy)
  3. Tandem HDCT/autoSCT
     * First HDCT (cyclophosphamide, etoposide, carboplatin)
     * Second HDCT (total body irradiation, thiotepa, melphalan)
  4. Local radiotherapy
  5. Retinoic acid, interleukin-2
  Interventions: Drug: Cyclophosphamide; Drug: Etoposide; Drug: Carboplatin; Drug: Thiotepa; Drug: Melphalan; Radiation: Total body irradiation

INTERVENTIONS:
Drug: Cyclophosphamide — First HDCT
Drug: Etoposide — First HDCT
Drug: Carboplatin — First HDCT
Drug: Thiotepa — Second HDCT
Drug: Melphalan — Second HDCT
Radiation: Total body irradiation — Second HDCT

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of tandem HDCT/ASCR in children with high-risk neuroblastoma. In the present study, a single arm trial of tandem HDCT/ASCR will be carried out. In the present study, the investigators will investigate whether tandem HDCT/ASCR might improve the survival of patients with high-risk neuroblastoma with acceptable toxicity.

DETAILED DESCRIPTION:
The prognosis of high-risk neuroblastoma after conventional chemoradiotherapy is generally poor. Therefore, a strategy using high-dose chemotherapy and autologous stem cell rescue (HDCT/ASCR) has been explored to improve the prognosis of patients with high-risk neuroblastoma. This strategy is based on the hypothesis that dose escalation might improve the survival of children with high-risk neuroblastoma. The results of randomized trials comparing HDCT/ASCR with chemotherapy alone showed a better event-free survival (EFS) in the HDCT/ASCR arm than in the continuous chemotherapy arm. However, the overall EFS was unsatisfactory.

In this context, investigators have examined the efficacy of double or triple tandem HDCT/ASCR to further improve the outcome of high-risk neuroblastoma patients. George et al. carried out a single arm trial of tandem transplantation as consolidation therapy, and reported improved long-term survival (5-year progression-free survival 47%) with acceptable toxicity. Kletzel et al. also conducted a single arm trial of triple tandem transplantation and reported improved survival (3-year EFS 57%). They demonstrated that further dose escalation using sequential HDCT/ASCR might result in further improvements in the survival of patients with high-risk neuroblastoma.

Investigators in the present study also carried out tandem transplantation as consolidation therapy, and reported improved long-term survival (5-year progression-free survival 62%) with acceptable toxicity. However, throughout our previous study, multiple modifications were made in the treatment plan, which resulted in significant variability over time between patients. This variability may create doubt as to whether tandem HDCT/ASCR itself resulted in the improved outcome. In addition, toxic death rate was relatively high (15.4%), although final survival rate was very high (best survival rate ever reported). Therefore, prospective study is needed to evaluate the efficacy and toxicity of tandem HDCT/ASCR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-risk neuroblastoma
* Patients with intermediate-risk neuroblastoma if gross tumor remained after surgery

Exclusion Criteria:

* Patients with progressive disease before high-dose chemotherapy
* Patients whose parents want to stop or change the planned treatment
* Patients with organ toxicities of NCI grade >2 before high-dose chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-08; Primary Completion 2015-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Overall survival and event-free survival, short-term and long-term toxicity of tandem high-dose chemotherapy and autologous stem cell transplantation | from 1 year after second high-dose chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Sung, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea